CLINICAL TRIAL: NCT00758043
Title: A Randomized Study of Stopping Treatment at 24 Weeks or Continuing Treatment to 48 Weeks in Treatment-Naïve Subjects With Genotype 1 Chronic Hepatitis C Who Achieve an Extended Rapid Viral Response While Receiving Telaprevir, Peginterferon Alfa2a (Pegasys®) and Ribavirin (Copegus®)
Brief Title: A Study Evaluating 24-Week and 48-Week Telaprevir-Based Regimen in Treatment Naïve Subjects With Genotype 1 Chronic Hepatitis C Who Achieve an Extended Rapid Viral Response
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Tibotec Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX08-950-111; EudraCT 2008-003836-39
Record Dates: First submitted 2008-09-19; First posted 2008-09-23 (Estimated); Results first posted 2011-07-21 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Hepatitis C
Keywords: Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- T12PR24 (eRVR+) (Experimental): Randomized Group: Telaprevir + Peg-IFN-alfa-2a + RBV for 12 weeks, followed by Peg-IFN-alfa-2a + RBV for 12 weeks; subjects achieved an extended rapid viral response (eRVR+) and were randomized to this group
  Interventions: Drug: telaprevir; Drug: ribavirin; Biological: peginterferon alfa-2a
- T12PR48 (eRVR+) (Experimental): Randomized Group: Telaprevir + Peg-IFN-alfa-2a + RBV for 12 weeks, followed by Peg-IFN-alfa-2a + RBV for 36 weeks; subjects achieved an extended rapid viral response (eRVR+) and were randomized to this group
  Interventions: Drug: telaprevir; Drug: ribavirin; Biological: peginterferon alfa-2a
- T12PR48 (eRVR-) (Experimental): Assigned Group: Telaprevir + Peg-IFN-alfa-2a + RBV for 12 weeks, followed by Peg-IFN-alfa-2a + RBV for 36 weeks; subjects did not achieve an extended rapid viral response and were assigned to this group
  Interventions: Drug: telaprevir; Drug: ribavirin; Biological: peginterferon alfa-2a
- Other (Experimental): Other Group: Subjects who received at least 1 dose of study drug, but prematurely discontinued treatment before Week 20, were not randomized or assigned to a treatment regimen.
  Interventions: Drug: telaprevir; Drug: ribavirin; Biological: peginterferon alfa-2a

INTERVENTIONS:
Drug: telaprevir — 750 mg every 8 hours (q8h) for 12 weeks
  Other Names: VX-950
Drug: ribavirin — 1000 - 1200 mg/day based on body weight for either 24 or 48 weeks
  Other Names: Copegus
Biological: peginterferon alfa-2a — 180 mcg/week for either 24 or 48 weeks
  Other Names: Pegasys

SUMMARY:
This study is being conducted to learn more about the safety and effect of telaprevir in combination with peginterferon alfa-2a (PEG-IFN) and ribavirin (RBV) in participants with hepatitis C who have never been treated for their hepatitis C virus (HCV). The study is designed to look at the relative benefits of 24 or 48 weeks of total treatment in people who respond quickly to a telaprevir-based treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has not received any previous treatment with any approved or investigational drug or drug regimen for the treatment of hepatitis C
* Male and female subjects, 18 to 70 years of age, inclusive
* Genotype 1, chronic hepatitis C with detectable HCV RNA.
* Screening laboratory values, tests, and physical exam within acceptable ranges
* Able and willing to follow contraception requirements
* Able to read and understand, and willing to sign the informed consent form and abide by the study restrictions.

Exclusion Criteria:

* Subject has any contraindications to Pegasys® or Copegus® therapy
* Evidence of hepatic decompensation in cirrhotic subjects
* History of organ transplant
* History of, or any current medical condition which could impact the safety of the subject in participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Adler, MD, PhD, Principal Investigator — Erasmus Hospital Bruxelles; Hendrik Reesink, MD, PhD, Principal Investigator — Academic Medical Center of the University of Amsterdam; Kenneth Sherman, MD, PhD, Principal Investigator — University of Cincinnati
Locations (66):
- United States (60):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Fresno, California
  - La Jolla, California
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - Aurora, Colorado
  - Farmington, Connecticut
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Marietta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Downers Grove, Illinois
  - Indianapolis, Indiana
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Hyattsville, Maryland
  - Laurel, Maryland
  - Boston, Massachusetts
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Novi, Michigan
  - Rochester, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Lebanon, New Hampshire
  - Atlantic City, New Jersey
  - Egg Harbor, New Jersey
  - Albuquerque, New Mexico
  - Bayside, New York
  - Manhasset, New York
  - New York, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Statesville, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Providence, Rhode Island
  - Columbia, South Carolina
  - Germantown, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Falls Church, Virginia
  - Seattle, Washington
  - Tacoma, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Belgium (3):
  - Brussels
  - Ghent
  - Liège
- Netherlands (2):
  - Amsterdam
  - Arnhem
- Santurce, Puerto Rico

REFERENCES:
- [Derived] Sherman KE, Flamm SL, Afdhal NH, Nelson DR, Sulkowski MS, Everson GT, Fried MW, Adler M, Reesink HW, Martin M, Sankoh AJ, Adda N, Kauffman RS, George S, Wright CI, Poordad F; ILLUMINATE Study Team. Response-guided telaprevir combination treatment for hepatitis C virus infection. N Engl J Med. 2011 Sep 15;365(11):1014-24. doi: 10.1056/NEJMoa1014463. PMID 21916639

RESULTS

PARTICIPANT FLOW:
Groups:
- T12PR24 (eRVR+): Telaprevir + peginterferon-alfa-2a (Peg-IFN-alfa-2a) + ribavirin (RBV) for 12 weeks, followed by 12 weeks of Peg-IFN-alfa-2a and RBV; subjects achieved an extended rapid viral response (eRVR+) and were randomized to this group
- T12PR48 (eRVR+): Telaprevir + Peg-IFN-alfa-2a + RBV for 12 weeks, followed by 36 weeks of Peg-IFN-alfa-2a and RBV; subjects achieved an extended rapid viral response (eRVR+) and were randomized to this group
- T12PR48 (eRVR-): Telaprevir + Peg-IFN-alfa-2a + RBV for 12 weeks, followed by 36 weeks of Peg-IFN-alfa-2a and RBV; subjects did not achieve an extended rapid viral response (eRVR-) and were assigned to this group
- Other: Subjects who received at least 1 dose of study drug, but prematurely discontinued treatment before Week 20 were not randomized or assigned to a treatment regimen.
Period: Overall Study
Arm/Group | T12PR24 (eRVR+) | T12PR48 (eRVR+) | T12PR48 (eRVR-) | Other
Started | 162 | 160 | 118 | 100
Completed | 161 | 119 | 79 | 0
Not Completed | 1 | 41 | 39 | 100
Not completed — Adverse Event | 1 | 20 | 12 | 62
Not completed — Lack of Efficacy | 0 | 6 | 18 | 12
Not completed — Refused Further Treatment | 0 | 11 | 5 | 8
Not completed — Lost to Follow-up | 0 | 2 | 2 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 4
Not completed — Required Prohibited Medication | 0 | 0 | 1 | 3
Not completed — Non-Compliant With study Drug | 0 | 0 | 0 | 1
Not completed — Other Reasons | 0 | 1 | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- T12PR24 (eRVR+): Telaprevir + Peg-IFN-alfa-2a + RBV for 12 weeks, followed by 12 weeks of Peg-IFN-alfa-2a and RBV; subjects achieved an extended rapid viral response (eRVR+) and were randomized to this group
- Total: Total of all reporting groups
Arm/Group | T12PR24 (eRVR+) | T12PR48 (eRVR+) | T12PR48 (eRVR-) | Other | Total
Number analyzed (Participants) | 162 | 160 | 118 | 100 | 540
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 158 | 157 | 118 | 99 | 532
  >=65 years | 4 | 3 | 0 | 1 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.6 (8.9) | 48.3 (9.9) | 49.5 (8.7) | 51.6 (8.4) | 49.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 63 | 48 | 46 | 215
  Male | 104 | 97 | 70 | 54 | 325
Region of Enrollment [Number; unit: participants]
  North America | 154 | 151 | 106 | 98 | 509
  Europe | 8 | 9 | 12 | 2 | 31

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Randomized Subjects Achieving Sustained Viral Response (SVR), Demonstrated by Achieving Undetectable HCV RNA 24 Weeks After Last Dose of Study Treatment (SVR24)
Description: SVR24planned was used to measure the primary outcome. SVR24 planned is defined as undetectable HCV RNA levels at the end of treatment (EOT) visit and at 24 weeks after the last planned dose of study treatment without any confirmed detectable HCV RNA levels in between those visits. All plasma HCV RNA levels were assessed using the Roche TaqMan HCV RNA assay (Version 2.0, lower limit of quantification [LLOQ] of 25 IU/mL).
Time Frame: 24 weeks after the last planned dose of study treatment
Population: The population analyzed included all subjects in the Full Analysis (FA) Set. All subjects in the FA Set received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | T12PR24 (eRVR+) | T12PR48 (eRVR+) | T12PR48 (eRVR-) | Other
Number analyzed (Participants) | 162 | 160 | 118 | 100
participants
  SVR24 (Statistical Analysis 1) | 149 | 140 | 76 | 23
  SVR24 (Statistical Analysis 2) | 149 | 144 | 78 | 27
Statistical Analysis 1: Comparison: T12PR24 (eRVR+) vs T12PR48 (eRVR+); Primary efficacy analysis was based on CI estimates (using the normal approximation, confidence limits were constructed for the difference in proportions) to rule out the inferiority of the T12/PR24/eRVR+ treatment regimen relative to the T12/PR48/eRVR+ treatment regimen. SVR24 was defined as undetectable HCV RNA at end of treatment through 24 weeks after the last planned dose; Test type: Non-Inferiority or Equivalence — Estimated by evaluating the treatment differences in the SVR24planned rates (T12PR24/eRVR+ minus T12PR48/eRVR+) and the 95% CI for these groups (the entire 2 sided CI is to the right of the predefined non-inferiority margin of -10.5%); Difference in proportions = 4.5, 95% CI 2-sided [-2.1 to 11.1]
Statistical Analysis 2: Comparison: T12PR24 (eRVR+) vs T12PR48 (eRVR+); SVR24 was defined as below the limit of quantitation at 24 weeks after the planned end of treatment. For subjects who had missing data at week 24 after the planned end of treatment, the week 12 data or the last follow-up time point after week 12 was carried forward for determining SVR24; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in proportions = 2.0, 95% CI 2-sided [-4.3 to 8.2]

2. Secondary Outcome: Proportion of Subjects Who Have Undetectable HCV RNA at Week 72
Description: SVR at Week 72 is defined as achieved SVR24planned and undetectable HCV RNA at Week 72 without any confirmed detectable HCV RNA levels in between those visits.
Time Frame: 72 weeks after the last planned dose of study treatment
Population: as for outcome 1
Measure: Number; unit: participants
Groups:
- T12PR24 (eRVR+): Telaprevir + Peg-IFN-alfa-2a + RBV for 12 weeks, followed by 12 weeks of Peg-IFN-alfa-2a and RBV; subjects achieved an extended rapid viral response and were randomized to this group
- T12PR48 (eRVR+): Telaprevir + Peg-IFN-alfa-2a + RBV for 12 weeks, followed by 36 weeks of Peg-IFN-alfa-2a and RBV; subjects achieved an extended rapid viral response and were randomized to this group
- T12PR48 (eRVR-): Telaprevir + Peg-IFN-alfa-2a + RBV for 12 weeks, followed by 36 weeks of Peg-IFN-alfa-2a and RBV; subjects did not achieve an extended rapid viral response and were assigned to this group (not randomized)
- Other: Subjects who received at least 1 dose of study drug, but prematurely discontinued treatment before Week 20, were not randomized or assigned to a treatment regimen
Arm/Group | T12PR24 (eRVR+) | T12PR48 (eRVR+) | T12PR48 (eRVR-) | Other
Number analyzed (Participants) | 162 | 160 | 118 | 100
participants | 141 | 140 | 76 | 20
Statistical Analysis 1: Comparison: T12PR24 (eRVR+) vs T12PR48 (eRVR+); Test type: Non-Inferiority or Equivalence — Estimated by evaluating the treatment differences in the SVR at Week 72 planned rates (T12PR24/eRVR+ minus T12PR48/eRVR+) and the 95% CI for these groups (the entire 2 sided CI is to the right of the predefined non-inferiority margin of 10.5%); Difference in Proportion = -0.5, 95% CI 2-sided [-7.7 to 6.8]
Statistical Analysis 2: Comparison: T12PR24 (eRVR+) vs T12PR48 (eRVR+); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Odds Ratio, log = 0.94, 95% CI 2-sided [0.49 to 1.82]

3. Secondary Outcome: Proportion of Subjects Achieving eRVR (Extended RVR), Demonstrated by Achieving Undetectable HCV RNA at Week 4 and at Week 12
Description: Extended rapid viral response is defined undetectable HCV RNA levels at Week 4 and Week 12 (on treatment).
Time Frame: Week 4 and Week 12
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | T12PR24 (eRVR+) | T12PR48 (eRVR+) | T12PR48 (eRVR-) | Other
Number analyzed (Participants) | 162 | 160 | 118 | 100
participants | 162 | 159 | 0 | 31

4. Secondary Outcome: Proportion of Randomized Subjects Who Have Undetectable HCV RNA 12 Weeks After Last Dose of Study Treatment
Description: SVR12 is defined as undetectable HCV RNA levels 12 weeks after the last planned dose of study treatment.
Time Frame: 12 weeks after last dose of study treatment
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | T12PR24 (eRVR+) | T12PR48 (eRVR+) | T12PR48 (eRVR-) | Other
Number analyzed (Participants) | 162 | 160 | 118 | 100
participants | 151 | 144 | 79 | 28

5. Secondary Outcome: Proportion of Subjects Who Have Undetectable HCV RNA at the EOT (Week 24 or Week 48 Respectively)
Time Frame: Week 24 or Week 48
Measure: Number; unit: participants
Arm/Group | T12PR24 (eRVR+) | T12PR48 (eRVR+) | T12PR48 (eRVR-) | Other
Number analyzed (Participants) | 162 | 160 | 118 | 100
participants | 159 | 154 | 97 | 59

6. Secondary Outcome: Proportion of Randomized Subjects Who Relapse
Description: Proportion of randomized subjects who relapsed was defined as the number of subjects who completed treatment, had undetectable HCV RNA at end of treatment (EOT; Week 24 or Week 48 respectively), and became HCV RNA detectable during antiviral follow-up (24 weeks after EOT).
Time Frame: From EOT to Week 48 or Week 72
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | T12PR24 (eRVR+) | T12PR48 (eRVR+) | T12PR48 (eRVR-) | Other
Number analyzed (Participants) | 162 | 160 | 118 | 100
participants | 9 | 1 | 5 | 0

7. Secondary Outcome: Proportion of Enrolled Subjects Who Relapse
Description: Proportion of enrolled subjects who relapsed was defined as the number of subjects who had undetectable HCV RNA at the EOT, and became HCV RNA detectable during antiviral follow-up.
Time Frame: From EOT to Week 48 or Week 72
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | T12PR24 (eRVR+) | T12PR48 (eRVR+) | T12PR48 (eRVR-) | Other
Number analyzed (Participants) | 162 | 160 | 118 | 100
participants | 9 | 4 | 11 | 13

8. Secondary Outcome: Safety and Tolerability as Assessed by Number of Subjects With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 72
Population: The population analyzed included all subjects who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | T12PR24 (eRVR+) | T12PR48 (eRVR+) | T12PR48 (eRVR-) | Other
Number analyzed (Participants) | 162 | 160 | 118 | 100
participants
  Subjects With AEs | 161 | 160 | 117 | 99
  Subjects With SAEs | 4 | 16 | 7 | 22

ADVERSE EVENTS:
Arm/Group | T12PR24 (eRVR+) | T12PR48 (eRVR+) | T12PR48 (eRVR-) | Other
Serious Adverse Events (participants affected / at risk) | 4/162 | 16/160 | 7/118 | 22/100
Other Adverse Events (participants affected / at risk) | 161/162 | 160/160 | 117/118 | 99/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T12PR24 (eRVR+) (N=162) | T12PR48 (eRVR+) (N=160) | T12PR48 (eRVR-) (N=118) | Other (N=100)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 4 | 0 | 7
ANAEMIA HAEMOLYTIC AUTOIMMUNE (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 2 | 1 | 0
APPENDICITIS (Infections and infestations) | 1 | 0 | 0 | 0
BACTERAEMIA (Infections and infestations) | 0 | 1 | 0 | 0
BACTERIAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
BURSITIS INFECTIVE (Infections and infestations) | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1 | 0
PNEUMONIA STAPHYLOCOCCAL (Infections and infestations) | 0 | 1 | 0 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 1
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 0 | 0 | 1
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 0 | 1 | 0 | 0
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
SPLENIC RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
CRYPTOGENIC ORGANISING PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 0 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1 | 0 | 0
PAPILLOEDEMA (Eye disorders) | 0 | 0 | 0 | 1
RETINOPATHY (Eye disorders) | 0 | 0 | 0 | 1
BILE DUCT STONE (Hepatobiliary disorders) | 0 | 1 | 0 | 0
LIVER DISORDER (Hepatobiliary disorders) | 0 | 0 | 0 | 1
BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
THROAT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
MANIA (Psychiatric disorders) | 0 | 0 | 1 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 0 | 0 | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 1
HAEMORRHAGIC ARTERIOVENOUS MALFORMATION (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 1 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 1 | 0
POLYMYOSITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
MIGRAINE (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T12PR24 (eRVR+) (N=162) | T12PR48 (eRVR+) (N=160) | T12PR48 (eRVR-) (N=118) | Other (N=100)
FATIGUE (General disorders) | 110 | 111 | 81 | 67
INFLUENZA LIKE ILLNESS (General disorders) | 47 | 40 | 33 | 21
CHILLS (Gastrointestinal disorders) | 30 | 39 | 19 | 26
PYREXIA (General disorders) | 20 | 32 | 22 | 22
IRRITABILITY (General disorders) | 30 | 26 | 24 | 12
INJECTION SITE ERYTHEMA (General disorders) | 23 | 23 | 18 | 17
PAIN (General disorders) | 14 | 18 | 6 | 9
OEDEMA PERIPHERAL (General disorders) | 7 | 11 | 4 | 1
INJECTION SITE RASH (General disorders) | 6 | 7 | 8 | 1
INJECTION SITE REACTION (General disorders) | 9 | 7 | 4 | 2
MALAISE (General disorders) | 1 | 9 | 1 | 2
PRURITUS (Skin and subcutaneous tissue disorders) | 95 | 83 | 55 | 40
RASH (Skin and subcutaneous tissue disorders) | 60 | 62 | 47 | 33
ALOPECIA (Skin and subcutaneous tissue disorders) | 28 | 49 | 33 | 6
DRY SKIN (Skin and subcutaneous tissue disorders) | 27 | 25 | 24 | 7
RASH MACULO-PAPULA (Skin and subcutaneous tissue disorders) | 27 | 17 | 11 | 6
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 19 | 19 | 10 | 9
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 10 | 9 | 9 | 8
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 9 | 12 | 5 | 4
RASH MACULAR (Skin and subcutaneous tissue disorders) | 8 | 6 | 5 | 7
ERYTHEMA (Skin and subcutaneous tissue disorders) | 8 | 8 | 4 | 2
NAUSEA (Gastrointestinal disorders) | 71 | 76 | 61 | 45
DIARRHOEA (Gastrointestinal disorders) | 48 | 54 | 38 | 24
VOMITING (Gastrointestinal disorders) | 25 | 26 | 25 | 20
ANORECTAL DISCOMFORT (Gastrointestinal disorders) | 35 | 25 | 18 | 8
HAEMORRHOIDS (Gastrointestinal disorders) | 29 | 23 | 15 | 11
DYSPEPSIA (Gastrointestinal disorders) | 18 | 21 | 13 | 8
CONSTIPATION (Gastrointestinal disorders) | 9 | 15 | 11 | 7
DRY MOUTH (Gastrointestinal disorders) | 10 | 13 | 12 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 9 | 12 | 8 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 10 | 12 | 4 | 2
ANAL PRURITUS (Gastrointestinal disorders) | 4 | 12 | 6 | 4
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 5 | 7 | 7 | 4
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 7 | 6 | 2 | 6
TOOTHACHE (Gastrointestinal disorders) | 2 | 5 | 7 | 0
HEADACHE (Nervous system disorders) | 61 | 57 | 51 | 35
DIZZINESS (Nervous system disorders) | 29 | 30 | 11 | 13
DYSGEUSIA (Nervous system disorders) | 18 | 24 | 14 | 6
DISTURBANCE IN ATTENTION (Nervous system disorders) | 5 | 11 | 9 | 4
HYPOAESTHESIA (Nervous system disorders) | 5 | 8 | 5 | 4
PARAESTHESIA (Nervous system disorders) | 3 | 8 | 6 | 1
INSOMNIA (Psychiatric disorders) | 50 | 62 | 44 | 26
DEPRESSION (Psychiatric disorders) | 22 | 35 | 28 | 22
ANXIETY (Psychiatric disorders) | 16 | 18 | 13 | 17
SLEEP DISORDER (Psychiatric disorders) | 1 | 2 | 6 | 0
ANAEMIA (Blood and lymphatic system disorders) | 68 | 66 | 38 | 40
NEUTROPENIA (Blood and lymphatic system disorders) | 23 | 36 | 31 | 13
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 4 | 6 | 6 | 5
LEUKOPENIA (Blood and lymphatic system disorders) | 4 | 6 | 6 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 34 | 41 | 37 | 15
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 30 | 40 | 19 | 18
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 13 | 12 | 17 | 7
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 10 | 9 | 10 | 9
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 7 | 9 | 5 | 5
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 2 | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 30 | 27 | 24 | 17
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 21 | 28 | 20 | 9
BACK PAIN (Musculoskeletal and connective tissue disorders) | 12 | 20 | 9 | 5
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 4 | 11 | 6 | 6
SINUSITIS (Infections and infestations) | 6 | 12 | 3 | 5
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 8 | 7 | 2
NASOPHARYNGITIS (Infections and infestations) | 6 | 4 | 7 | 1
BRONCHITIS (Infections and infestations) | 3 | 6 | 3 | 5
URINARY TRACT INFECTION (Infections and infestations) | 5 | 8 | 3 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 16 | 24 | 5 | 8
ANOREXIA (Metabolism and nutrition disorders) | 9 | 12 | 12 | 10
HYPOKALAEMIA (Metabolism and nutrition disorders) | 6 | 7 | 7 | 3
VISION BLURRED (Eye disorders) | 16 | 14 | 12 | 12
DRY EYE (Eye disorders) | 10 | 11 | 5 | 1
WEIGHT DECREASED (Investigations) | 7 | 15 | 9 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days